CLINICAL TRIAL: NCT04384744
Title: To Explore the Effect of Growth Hormone on Outcomes of in Vitro Fertilisation and Telomerase Activity of Granulosa Cells in Women With Poor Ovarian Response
Brief Title: To Explore the Effect of GH on Outcomes of IVF and Telomerase Activity of Granulosa Cells in Women With POR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019001
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-04

CONDITIONS: GH; Poor Ovarian Reserve Based on POSEIDON
Keywords: growth hormone; POSEIDON; low ovarian reserve; prospective observational cohort study
MeSH Terms: interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — follicular fluid abandoned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- GH-POR: Participants diagnosed POR according to POSEIDON criteria with low ovarian reserve undergo IVF in our center with long protocol or antagonist protocol and is adjuvant with GH 2IU/d from previous menstrual period for about six weeks.
  Interventions: Drug: growth hormone
- NGH-POR: Participants diagnosed POR according to POSEIDON criteria with low reserve undergo IVF in our center with long protocol or antagonist protocol without GH adjuvant.
- NGH-NOR: Participants with normal ovarian reserve undergo IVF in our center with long protocol or antagonist protocol without GH adjuvant.

INTERVENTIONS:
Drug: growth hormone — growth hormone was adjuvanted 2IU/d from previous menstrual period for about six weeks.
  Groups: GH-POR

SUMMARY:
It is still a big difficult clinical problem for patients with poor ovarian reserve undergoing in vitro fertilization. The decrease in both quality and quantity of egg are the main cause for poor clinical prognosis. Growth hormone (GH) is currently one of the main adjuvant for improving pregnancy outcomes in patients with POR, and the investigators' previous retrospective study suggested GH was effective in live birth rate in subgroup of patients with POR older than 35 years old. To further figure out the mechanism of GH effectiveness in POR patients and the effect on clinical outcomes in POR patients, the investigators designed this prospective observational cohort study.

ELIGIBILITY:
Inclusion Criteria:

For patients with poor ovarian response, the criteria is based on POSEIDON criteria[1]:

1. low ovarian reserve(AMH <1.2ng/ml, or AFC <5);
2. younger than 40.

For patients with normal ovarian reserve, the criteria is as follow:

1. Patients who are between 20-40 years old;
2. clinical diagnosis of non-functional fallopian tube;
3. regular menstrual cycles.

Exclusion Criteria:

1. BMI ≥28kg/m2;
2. medical diseases such as endocrine and metabolic diseases, autoimmune disease, etc;
3. ovarian neoplasm that ≥4 cm in diameter and has no clear pathological diagnosis by surgery;
4. adenomyosis or endometriosis confirmed by surgery;
5. untreated abnormal intrauterine environment, such as uterine effusion, endometritis, etc;
6. untreated hydrosalpinx;
7. polycystic ovary syndrome.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes patients diagnosed as POR based on POSEIDON criteria and with low ovairan reserve, as well as patients with normal ovairan reserve seeking for ART help due to pelvic tubal factors.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05-26 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 1-2 years
  Clinical pregnancy means pregnancy sac is seen intrauterine under ultrasound 7 weeks after embryo transferred.

SECONDARY OUTCOMES:
live birth rate | 1-2 years
  Live birth rate(%): number of live birth/ transferred cycle.
number of oocytes retrieved | 1-2 years
  number of oocytes retrieved on day of OPU

OTHER OUTCOMES:
telomerase activity of granulosa cells | 1-2 years
  detection of telomerase activity of granulosa cells in wasted follicular fluid

CONTACTS AND LOCATIONS:
Overall Officials: meihong Cai, master, Study Director — Guangzhou First People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622